CLINICAL TRIAL: NCT07011303
Title: Investigation of the Effect of Horizontal Platelet Rich Fibrin Placed in Tooth Extraction Sockets on Bone Formation
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Tokat Gaziosmanpasa University (Other)
Responsible Party: Principal Investigator, esengul sen, Dr. faculty member, Tokat Gaziosmanpasa University
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Prevention
Other Study IDs: 23-KAEK-320; 2024/25 (Other Grant/Funding Number: Tokat Gaziosmanpasa University Scientific Research Fund)
Record Dates: First submitted 2024-12-12; First posted 2025-06-08 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Tooth Loss; Dental Implant Failed; Alveolar Bone Loss
Keywords: H-PRF, L-PRF, tooth extraction
MeSH Terms: conditions — Tooth Loss; Alveolar Bone Loss

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- CONTROL GROUP (No Intervention): Control Group (n=10): Patient group in which no material was placed in the extraction socket after tooth extraction.
- L-PRF (leukocyte-platelet rich fibrin) (Active Comparator): L-PRF (Comparison Arm): The patient group in which L-PRF will be placed in the extraction socket after tooth extraction.
  Interventions: Procedure: L-PRF
- H-PRF (horizontal-platelet rich fibrin) (Experimental): H-PRF (Research Branch): The patient group in which H-PRF will be placed in the extraction socket after tooth extraction.
  Interventions: Procedure: H-PRF

INTERVENTIONS:
Procedure: H-PRF — Blood will be taken from the patient before the surgical procedure is started. The blood sample will be placed in the H-TZF device for centrifugation and the sample will be horizontally centrifuged (2200 RPMx8 min, 700g). After the blood is processed for centrifugation, the surgery will begin. Surgery will be performed under local anesthesia with articaine 2 ml 4% and epinephrine 1:100,000. All patients will be operated by the same surgeon. After local anesthesia is achieved, tooth extraction will be started. After tooth extraction, the surgical field will be washed with sterile 0.9% saline, and H-PRF material will be placed in the area and primarily sutured with a 3.0 silk suture. All patients will be given postoperative instructions by the surgeon. Patients will be prescribed mouthwash (0.12% chlorhexidine mouthwash twice daily for 7 days).
  Arms: H-PRF (horizontal-platelet rich fibrin)
Procedure: L-PRF — Blood will be taken from the patient before the surgical procedure is started. The blood sample will be placed in the L-PRF device for centrifugation and the sample will be centrifuged. (2700M x 12 min, 700g) After the blood is processed for centrifugation, the surgery will begin. Surgery will be performed under local anaesthesia with articaine 2 ml 4% and epinephrine 1:100,000. All patients will be operated by the same surgeon. After local anaesthesia is achieved, tooth extraction will be started. After tooth extraction, the surgical field will be washed with sterile 0.9% saline, and L-PRF material will be placed in the area and primarily sutured with a 3.0 silk suture. All patients will be given postoperative instructions by the surgeon. Patients will be prescribed mouthwash (0.12% chlorhexidine mouthwash twice daily for 7 days).
  Arms: L-PRF (leukocyte-platelet rich fibrin)

SUMMARY:
Dental implants, the treatment of complete and partial edentulous cases involving the restoration of lost teeth, have become a registered and widely used treatment option. Implants: It is an ideal option for the good oral health of the person who has lost his teeth due to periodontal disease, caries, trauma, or any other reason. When teeth are missing, melting occurs in the jawbone. Following tooth extraction, the loss of the implant and the amount of melting are significantly reduced.

In implant treatments, which have become widely used today, successful results depend on the ideal volume and quality of hard and soft tissues. The amount of bone present in the edentulous area is important for the indication of the implant.

The aim of this study is to evaluate the histological and immunohistochemical contribution of the H-PRF (horizontal-platelet rich fibrin) material placed in the extraction sockets to the quality of the newly formed bone tissue in order to make successful implants after tooth extractions for various reasons in humans.

The research hypothesis is that H-PRF will contribute positively to the healing of tooth extraction sockets.

DETAILED DESCRIPTION:
This study was planned as a prospective, randomized controlled, single-blind clinical study. The study will be conducted on patients applying to the Tokat Gaziosmanpasa University Faculty of Dentistry Oral and Maxillofacial Surgery clinic in the same clinic.

Study inclusion criteria: Volunteer ASA I individuals between the ages of 18-40

Exclusion criteria for the study: Those who are pregnant or lactating Those receiving anticoagulant or antiplatelet drug therapy Those who received radiotherapy to the head and face area Those who are allergic to local anesthetics and prescribed medications

Considering possible losses, a total of 30 volunteers will be included in the study.

Randomization: Before the operation, patients will be divided into three groups: a control group, an L-PRF (leukocyte platelet-rich fibrin) group, and an H-PRF group. The sealed envelope method will be used in the process of assigning patients to the group. Sealed envelopes of the same color will be used for each group, and the patient will not know which group he is assigned to, but the physician will know which group the patient is assigned to.

Tooth extraction will be performed on patients in each group. CBCT (cone beam computed tomography) will be taken immediately afterwards. Soft tissue healing will be evaluated in the first 7 days. CBCT will be taken again after 3 months. Dental implant operations will be performed. Bone tissue biopsies will be taken after the operation. Biopsies are not routine procedures and will be obtained from bone tissue that will be removed during the operation.

Control Group (n=10): Patient group in which no material was placed in the extraction socket after tooth extraction. There will be 10 patients in this group.

L-PRF (Comparison Arm): The patient group in which L-PRF will be placed in the extraction socket after tooth extraction. There will be 10 patients in this group. Patients will be called on the 2nd and 7th days, and their conditions will be evaluated.

H-PRF (Research Branch): The patient group in which H-PRF will be placed in the extraction socket after tooth extraction. There will be 10 patients in this group. Patients will be called on the 2nd and 7th days and their conditions will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Volunteer ASA I individuals between the ages of 18-40
* Individuals with indication for tooth extraction
* Patients who want to have implants after tooth extraction

Exclusion Criteria:

* Those who are pregnant or lactating
* Those receiving anticoagulant or antiplatelet drug therapy
* Those who received radiotherapy to the head and face area

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-06-01 (Actual); Primary Completion 2024-11-01 (Actual); Study Completion 2026-04-01 (Estimated)

PRIMARY OUTCOMES:
Maximum mouth opening measurements | Preoperative, postoperative 2nd day and 7th day
  Preoperative and postoperative maximum mouth opening will be measured between the lower and upper middle incisal teeth.
Pain level after extraction postoperative pain after tooth extraction | After 6th hour and 7th day (6th hour, 2nd day, 3rd day, 4th day, 5th day, 6th day, 7th day)
  Visual Analog Scale (VAS) will be used to assess pain.
Swelling | Postoperative 2nd and 7th days
  Preoperative and postoperative edema will be measured according to the reference points.

CONTACTS AND LOCATIONS:
Locations (1):
- Tokat Gaziosmanpasa University, Faculty of Dentistry, Tokat Province, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No